CLINICAL TRIAL: NCT06832319
Title: EFFECT of PERSONALIZED FEEDBACK USED in SIMULATION TECHNIQUE on KNOWLEDGE and SKILLS in MANAGEMENT of BLEEDING DURING PREGNANCY
Brief Title: IMPACT of KNOWLEDGE and SKILLS in MANAGEMENT of BLEEDING DURING PREGNANCY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, principal investigator_PhD midwife, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Burdur_Mehmet Akif Ersoy Uni
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bleeding Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- INTERVENTION 1 (Active Comparator)
  Interventions: Behavioral: PERSONALIZED FEEDBACK

INTERVENTIONS:
Behavioral: PERSONALIZED FEEDBACK — Students in the study group will be asked to intervene in a simulated situation in the management of bleeding during pregnancy. It will be filmed with a camera so that students can see their own mistakes after the simulated scenario. After the scenarios are completed by the students in the control group, the mistakes in the clinical situations will be analyzed by the researchers and students in the form of questions and answers and the necessary feedback will be given to them.
  Arms: INTERVENTION 1

SUMMARY:
Simulation training motivates participants to interact and collaborate, and studies on interdisciplinary groups show that it improves soft skills such as communication and teamwork. Midwifery students' skills are the ability to apply knowledge and use their knowledge to perform tasks and solve problems. They are cognitive in nature and include logical, intuitive and creative thinking. Practical experiences such as the application of skills and methods, materials, tools and equipment further develop these skills. Skills represent the application of learned abilities and the result of practical experience that emerges both cognitively and practically. In addition, feedback is included in the methods used as an important part of clinical education

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research, Continuing their sophomore year in the 2024-2025 Spring semester,

Exclusion Criteria:

* Students who do not participate in theoretical explanation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Scale for Evaluating Simulation-Based Learning | 1 HOUR
Student Satisfaction and Self-Confidence Scale in Learning | 1 HOUR